CLINICAL TRIAL: NCT01992588
Title: A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of FIAsp When Administered as a Bolus in a Continuous Subcutaneous Infusion Regimen in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3890; 2011-000913-37 (EudraCT Number); U1111-1119-5358 (Other: WHO)
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp followed by NovoRapid® (Experimental): Each subject will be randomly allocated to a treatment sequence consisting of 2 dosing visits separated by a wash-out period of 3-12 days
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® followed by FIAsp (Experimental): Each subject will be randomly allocated to a treatment sequence consisting of 2 dosing visits separated by a wash-out period of 3-12 days
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Subjects - in a euglycaemic clamp setting - will receive a priming (initial) dose followed by a continuous basal rate infusion and finally a bolus dose on top of the basal rate infusion.
  The trial products will be administered subcutaneously (s.c. under the skin) by means of an insulin pump.
  Arms: FIAsp followed by NovoRapid®
Drug: insulin aspart — Subjects - in a euglycaemic clamp setting - will receive a priming (initial) dose followed by a continuous basal rate infusion and finally a bolus dose on top of the basal rate infusion.
  The trial products will be administered subcutaneously (s.c. under the skin) by means of an insulin pump.
  Arms: NovoRapid® followed by FIAsp

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to compare the pharmacokinetic (the exposure of the trial drug in the body) and pharmacodynamic (the effect of the investigated drug on the body) properties of FIAsp (faster-acting insulin aspart) and insulin aspart (NovoRapid®) given as a bolus on top of a basal continuous subcutaneous insulin infusion (CSII).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-64 years (both inclusive) at the time of signing informed consent
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index (BMI) 18.5-28.0 kg/m^2 (both inclusive)
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for at least 12 months

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
CSII bolus related baseline corrected area under the serum insulin aspart concentration-time curve | From 0 to 30 minutes

SECONDARY OUTCOMES:
CSII bolus related baseline corrected area under the serum insulin aspart concentration-time curve | From 0 to 1 hour
CSII bolus related baseline corrected area under the glucose infusion rate curve | From 0 to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Zijlstra E, Nosek L, Rikte T, Haahr H. Pharmacological properties of faster-acting insulin aspart vs insulin aspart in patients with type 1 diabetes receiving continuous subcutaneous insulin infusion: A randomized, double-blind, crossover trial. Diabetes Obes Metab. 2017 Feb;19(2):208-215. doi: 10.1111/dom.12803. Epub 2016 Nov 14. PMID 27709762
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com